CLINICAL TRIAL: NCT02742792
Title: Effect of Strength Training on Sleep Apnea in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0613
Record Dates: First submitted 2016-04-01; First posted 2016-04-19 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; elderly; exercise
MeSH Terms: conditions — Sleep Apnea Syndromes; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): Resistance training, twice a week during 12 weeks.
  Interventions: Other: Resistance training
- Advice on lifestyle (Other): Patients receive advice on lifestyle. Patients will be asked to participate in the elderly group meetings the basic health unit linked to the hospital.
  Interventions: Other: Advice on Lifestyle

INTERVENTIONS:
Other: Resistance training — Twenty-four strength training sessions consisted in exercises of extension and flexion knees, lat pull-down, elbow extension and flexion, sitting bench press and hip abduction.
  Arms: Resistance training
Other: Advice on Lifestyle — Patients receive advice on lifestyle. Patients will be asked to participate in the elderly group meetings the basic health unit linked to the hospital.
  Arms: Advice on lifestyle

SUMMARY:
The objective of the study is to evaluate the impact of strength training on sleep apneas in the elderly. Individuals aged between 65 and 80 years and that presenting apnea-hypopnea index between 20 and 50 events per hour, measured by out-of-center portable polysomnography, will be recruited. Those included will be randomized to two groups: Intervention: consisted of 12 weeks, twice a week, of strength training; or control: consisted of lifestyle recommendations.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a disorder that exposes the individual to repeated periods of hypoxia and awakenings during sleep. OSA occurs in up to one third of the population, constituting a public health problem. The prevalence of sleep apnea increases with age, reaching up to 90%. Its consequences include sympathetic nervous system activation, increased blood pressure and heart rate, myocardial contractility overload, decline in parasympathetic activity, oxidative stress, systemic inflammation, platelet activation, and impaired vascular endothelial function. OSA is a risk factor for hypertension, coronary artery disease, peripheral artery disease, heart failure, and arrhythmias. The classical treatment options for OSA are the use of continuous positive airway pressure, oral appliances for mandibular advancement, surgery, weight reduction, and lifestyle change, including recommendation of regular practice of exercise.

Physical exercise is accepted culturally and scientifically as a non-pharmacological intervention beneficial to health. Aerobic and resistance exercises improve the quality of sleep. There is evidence of improvement in the general well-being and, particularly in sleep. Promote or improve sleep through exercise is healthy, safe, and simple. A sedentary lifestyle is linked with a higher incidence and severity of sleep apnea. Increase in the number of hours of exercise reduces these problems. Exercise has been used with consistent results to treat OSA. The effect size of exercise in treatment of OSA ranges between 0.4 and 1.5 standard deviations. In a meta-analysis, totaling 129 participants, the mean effect was the reduction of 7 events per hour. Although the results of randomized clinical trials and other studies pointing to the decrease in AHI after physical training, all studies involved adult populations with an average age between 42 and 54 years. The role of exercise in the elderly with OSA, the most affected population, remains uninvestigated.

The research question is: What is the effect of strength training on the apnea-hypopnea index (AHI) in elderly with OSA? The objective of the study is to evaluate the impact of strength training on OSA in the elderly.

The trial will recruit individuals aged 65 to 80 years ascribed to a primary care unit linked to the university hospital. Individuals that accept to participate in the study, will undergo out-of-center polysomnography in order to detect and quantify the severity of OSA. Individuals with AHI between 20 and 50 events per hour will be eligible, and will be randomly allocated to the intervention or the control group. Randomization will be performed by sequence numbers generated by computer at randomization.com.

Individuals allocated to the intervention group will hold two sessions per week of strength training consisted of exercises for legs, arms, chest, back, and abdomen in the university Physical Education High School, during 12 weeks. The individuals allocated to the control group will receive advice on lifestyle and will participate in the meetings of an elderly social group in the basic health unit. All individuals from both groups will perform an evaluation consisting of body composition by bioelectrical impedance, maximum dynamic force by 1-repetition maximum strength test, quality and muscle thickness by ultrasound, and physical function by Sit-to-stand test, Timed up and go test and Handgrip strength test. All evaluations will be repeated at the end of the 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 80 years
* Both genders
* Not being engaged in regular structured resistance exercise
* Apnea-hypopnea index between 20 and 50 events per hour
* Time availability to include physical activity in routine
* Consenting to participate in the survey

Exclusion Criteria:

* Being in treatment for sleep apnea
* Osteoarticular problems that compromise the exercises included in the project
* Neuromuscular Problems
* Serious illness
* Uncontrolled hypertension
* Acute myocardial infarction in the last year
* Recent trauma of the upper airway
* Other chronic diseases in treatment for over a month in the last year
* Drugs with effect on the central nervous system

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 12 weeks
  Measured by out-of-center polysomnography

SECONDARY OUTCOMES:
Muscle strength | 12 weeks
  Measured by 1-repetition maximum strength test
Muscle thickness | 12 weeks
  Measured by ultrasound
Muscle quality | 12 weeks
  Measured by ultrasound
Muscle strength of legs | 12 weeks
  Measured by Sit-to-stand test
Mobility | 12 weeks
  Measured by Timed up and go test
Grip strength | 12 weeks
  Measured by Handgrip strength test

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martinez, PhD, Principal Investigator — Graduate Program in Cardiology and Cardiovascular Sciences, Universidade Federal do Rio Grande do Sul (UFRGS), Porto Alegre, RS, Brazil; Cardiology Unit, Hospital de Clinicas de Porto Alegre (HCPA - UFRGS), Porto Alegre, RS, Brazil
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] da Silva RP, Martinez D, Uribe Ramos JM, Martins EF, Tedesco-Silva LM, Lopez P, Cadore EL. The effects of resistance exercise on obstructive sleep apnea severity and body water content in older adults: A randomized controlled trial. Sleep Med. 2022 Jul;95:37-46. doi: 10.1016/j.sleep.2022.04.014. Epub 2022 Apr 22. PMID 35561473
- [Derived] da Silva RP, Martinez D, Lopez P, Cadore EL. Effect of strength training on sleep apnea severity in the elderly: study protocol for a randomized controlled trial. Trials. 2017 Oct 23;18(1):489. doi: 10.1186/s13063-017-2238-3. PMID 29058628